CLINICAL TRIAL: NCT06166719
Title: Prediction of Complications After Major Gastrointestinal Surgery With Machine Learning and Point of Care Ultrasound: an Observational Cohort Study.
Brief Title: Prediction of Complications After Major Gastrointestinal Surgery With Machine Learning and Point of Care Ultrasound
Acronym: AI_PLUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, A.P.J. Vlaar, prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL84107.018.23
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Surgery-Complications; Overload Fluid
Keywords: Intensive care unit; Gastro-intestinal surgery; Prediction
MeSH Terms: conditions — Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peri-operative blood samples for hormone levels and liver metabolism e.g. Whole blood and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This is an observational study in patients undergoing major surgery. In which we attempt to predict complications (e.g. low blood pressure, ICU-admittance after major surgery using continuous blood pressure measurements. We will also attempt to predict their response to fluid therapy using point of care ultrasound. Eventually we aim to combine these methods to detect complications earlier and to give advice about whether or not administration of fluid is appropriate

DETAILED DESCRIPTION:
The primary aim of this study is to develop a machine learning framework to predict major complications after major gastro-intestinal surgery. Secondary aims include combining this framework with point of care ultrasound to determine the best initial resuscitative strategy; and to determine which ultrasound parameters are best predictive of fluid intolerance. Furthermore if the renin angiotensin aldosterone system is more active after liver resection.

Study design:

Single centre observational cohort study

Study population:

Adult patients undergoing elective major gastrointestinal surgery

Primary study parameters/outcome of the study:

The main study endpoint is a machine learning framework based on the hemodynamic profile to predict major complications,especially cardiovascular/pulmonary instability, including, sepsis and septic shock. Data from the ClearSight will be used to collect non-invasive arterial pressure waveforms. point of care ultrasound of heart, lungs and abdominal veins, and clinical data from the electronic medical record will be collected

Secondary study parameters/outcome of the study (if applicable):

point of care ultrasound of heart, lungs and abdominal veins, and clinical data from the electronic medical record will be collected. Ina subgroup of 40 patients RAAS levels and portal blood samples will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age.
* elective major gastrointestinal surgery: esophagectomy, gastrectomy, pancreatomy or major liver resection (3 segments or more).

Exclusion Criteria:

* no informed consent
* Patients with major cardiac shunts
* Patients with dialysis shunts or peritoneal dialysis
* Patients in whom POCUS is not possible or assessment of fluid status is unreliable e.g. BMI> 40, pulmonary fibrosis.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients who will undergo elective, major gastrointestinal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Post-operative complications | 28 days
  mainly complications such as ICU admission, re-OR, hemodynamic or respiratory instability, death, organ failure

SECONDARY OUTCOMES:
fluid overload or fluid intolerance | 28 days
  ultrasound measurements such as lung ultrasound and VExUS

OTHER OUTCOMES:
renin en aldosterone activity | 28 days
  pre and post-opative (day 0 day 1 and day 3) Renin and aldosterone levels in the blood

CONTACTS AND LOCATIONS:
Overall Officials: A.P. J. Vlaar, PhD, Principal Investigator — Department of Intensive Care, Amsterdam UMC
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
As of this moment it is undecided whether or not the individual patient data will be made available